CLINICAL TRIAL: NCT02163291
Title: Phase II Study of Paclitaxel Liposome Plus S-1 as Neoadjuvant Chemotherapy for Advanced Gastric Cancer
Brief Title: Study on Neoadjuvant Chemotherapy for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jiafu Ji, President, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS-01-2013
Record Dates: First submitted 2014-06-07; First posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Advanced Gastric Carcinoma
Keywords: advanced gastric cancer; neoadjuvant chemotherapy; safety; feasibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- paclitaxel liposome (Experimental): S-1 plus paclitaxel liposome
  Interventions: Drug: paclitaxel liposome

INTERVENTIONS:
Drug: paclitaxel liposome — S-1 40 mg/m2 bid d1-14 po and paclitaxel liposome 175mg/m2 d1 intravenously infusion for 3 hours, every 3 weeks. After 2 cycles' treatment, if clinical response is complete response（CR）,partial regression（PR） or stable disease（SD）, another 2 cycles is administered and operation is performed after the total 4 cycles. If response is progressive disease（PD）, chemotherapy is stopped and operation is performed.

SUMMARY:
Gastric cancer is the second cause of cancer related death and China has the most gastric cancer patients in the world. Although systemic strategies, including adjuvant chemotherapy, postoperative chemoradiotherapy, perioperative chemotherapy, have evolved and showed benefits these years, the prognosis of advanced gastric cancer is still not satisfactory. Optimal regimens and optimal method administration is still being found. Neoadjuvant chemotherapy has many advantages, including downstaging the tumor, increasing R0 rate, early eradicating of micrometastasis. In previous trials, combination of paclitaxel and s-1 has showed safety and tolerance in recurrent or metastatic gastric cancer. Using liposome as a carrier, paclitaxel has a better histocompatibility and cellular affinity, resulting a improved stability and reduced toxicity. In this phase II trial, we are going to study the safety and feasibility of paclitaxel liposome plus s-1 as neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric cancer
* Disease at clinical stage of resectable or potentially resectable(T3-4, N0-3, M0) by CT and endoscopic ultrasonography (EUS)
* Karnofsky performance status(KPS） ≥ 70
* No prior antitumor treatment is allowed, including chemotherapy, radiotherapy, immune therapy or target therapy
* Life expectancy more than 3 months
* Adequate organ function as defined below:White Blood Cell Count （WBC） ≥ 3.0*10^9/l, Absolute Neutrophil Count （ANC） ≥ 1.5*10^9/l, Hemoglobin ≥ 100 g/l, Platelets ≥ 100*10^9/l, Total Bilirubin （TBIL） ≤ 1.5mg/dl, Aspartate Aminotransferase（AST） and Alanine Aminotransferase(ALT) ≤ 2.5×ULN, Alkaline pPosphatase( ALP) ≤ 2.5×ULN, Renal Serum Creatinine < 1.5mg/dl
* Adequate lung and heart function

Exclusion Criteria:

* ≥ grade 2 neuropathy
* History of malignancy
* With uncontrolled central nervous system metastasis
* Concurrent disease or condition that would interfere with the subject's safety (including current active hepatic, biliary, renal, respiratory disease, acute infection, severe malnutrition, uncontrolled diabetes hypertension et al)
* Severely inadequate intake of water or diet

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | up to 24 weeks
  Pathology is usually reported 1 week after operation.The result of Pathological complete response rate will be accessed after all of the 30 participants operated.

SECONDARY OUTCOMES:
Object Response Rate | up to 24 weeks
  Object Response Rate(ORR) is defined as the percentage of CR and PR among all of the participants under best overall outcome evaluation .Pathology is usually reported 1 week after operation.The result of Object Response Rate will be accessed after all of the 30 participants operated.
Disease Control Rate | up to 24 weeks
  Disease Control Rate(DC R) is defined as the percentage of CR+PR+SD among all of the participants under best overall outcome evaluation .Pathology is usually reported 1 week after operation.The result of Disease Control Rate will be accessed after all of the 30 participants operated.
Number of Participants with Adverse Eventss a Measure of Safety and Tolerability | up to 12 weeks
  Participants will be followed during all the s a Measure of Safety and Tolerability4 circles of chemotherapy ,an expected average of 12 weeks.Number of participants with Adverse Events will calculated as a Measure of Safety and Tolerability.
R0 rate, surgical morbidity and mortality | 2 weeks
  The results of R0 rate, surgical morbidity and mortality will be accessed after operation ,participants will be followed for the duration of hospital stay, an expected average of 2 weeks .

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Haidian District, Beijing, China

REFERENCES:
- [Background] Wang X, Zhou J, Wang Y, Zhu Z, Lu Y, Wei Y, Chen L. A phase I clinical and pharmacokinetic study of paclitaxel liposome infused in non-small cell lung cancer patients with malignant pleural effusions. Eur J Cancer. 2010 May;46(8):1474-80. doi: 10.1016/j.ejca.2010.02.002. Epub 2010 Mar 6. PMID 20207133
- [Background] Zhang Q, Huang XE, Gao LL. A clinical study on the premedication of paclitaxel liposome in the treatment of solid tumors. Biomed Pharmacother. 2009 Sep;63(8):603-7. doi: 10.1016/j.biopha.2008.10.001. Epub 2008 Oct 31. PMID 19019625
- [Background] Chen L, Chen Q, Zhuang Z, Zhang Y, Tao J, Shen L, Shen X, Chen Z, Wang J, Zhu M, Wang H. Effect of the weekly administration of liposome-Paclitaxel combined with s-1 on advanced gastric cancer. Jpn J Clin Oncol. 2014 Mar;44(3):208-13. doi: 10.1093/jjco/hyt212. Epub 2014 Jan 22. PMID 24453274
- [Background] Huang D, Ba Y, Xiong J, Xu N, Yan Z, Zhuang Z, Yu Z, Wan H, Zhang Y, Deng T, Zheng R, Guo Z, Hu C, Wang M, Yu Z, Yao Y, Meng J. A multicentre randomised trial comparing weekly paclitaxel + S-1 with weekly paclitaxel + 5-fluorouracil for patients with advanced gastric cancer. Eur J Cancer. 2013 Sep;49(14):2995-3002. doi: 10.1016/j.ejca.2013.05.021. Epub 2013 Jun 27. PMID 23810466
- [Background] Lee JJ, Kim SY, Chung HC, Lee KH, Song HS, Kang WK, Hong YS, Choi IS, Lee YY, Woo IS, Choi JH. A multi-center phase II study of S-1 plus paclitaxel as first-line therapy for patients with advanced or recurrent unresectable gastric cancer. Cancer Chemother Pharmacol. 2009 May;63(6):1083-90. doi: 10.1007/s00280-008-0818-3. Epub 2008 Sep 24. PMID 18813927
- [Background] Nakajo A, Hokita S, Ishigami S, Miyazono F, Etoh T, Hamanoue M, Maenohara S, Iwashita T, Komatsu H, Satoh K, Aridome K, Morita S, Natsugoe S, Takiuchi H, Nakano S, Maehara Y, Sakamoto J, Aikou T; Kyushu Taxol TS-1 Study Group. A multicenter phase II study of biweekly paclitaxel and S-1 combination chemotherapy for unresectable or recurrent gastric cancer. Cancer Chemother Pharmacol. 2008 Nov;62(6):1103-9. doi: 10.1007/s00280-008-0693-y. Epub 2008 Mar 4. PMID 18317763
- [Background] Mochiki E, Ogata K, Ohno T, Toyomasu Y, Haga N, Fukai Y, Aihara R, Ando H, Uchida N, Asao T, Kuwano H; North Kanto Gastric Cancer Study Group. Phase II multi-institutional prospective randomised trial comparing S-1+paclitaxel with S-1+cisplatin in patients with unresectable and/or recurrent advanced gastric cancer. Br J Cancer. 2012 Jun 26;107(1):31-6. doi: 10.1038/bjc.2012.222. Epub 2012 May 22. PMID 22617130